CLINICAL TRIAL: NCT01871987
Title: Pharmacokinetic Study of FK949E -A Pharmacokinetic Study in Healthy Male Volunteers to Investigate the Effect of Food on the Pharmacokinetics of FK949E
Brief Title: Study to Evaluate the Effect of Food Intake on the Plasma Concentration Changes of Quetiapine After Oral Administration of FK949E in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 6949-CL-0003
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Healthy; Plasma Concentration Change of Quetiapine
Keywords: FK949E; Quetiapine; Antipsychotic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- fasted group (Experimental): receiving FK949E in fasted condition
  Interventions: Drug: FK949E
- low fat group (Experimental): receiving FK949E after low fat meal
  Interventions: Drug: FK949E
- high fat group (Experimental): receiving FK949E after high fat meal
  Interventions: Drug: FK949E

INTERVENTIONS:
Drug: FK949E — oral
  Other Names: extended release formulation of quetiapine

SUMMARY:
A study to evaluate the effect of food on the plasma concentration changes of quetiapine after oral administration of FK949E (extended release formulation of quetiapine) in healthy male subjects.

DETAILED DESCRIPTION:
This is a 3-way cross-over study.

ELIGIBILITY:
Inclusion Criteria:

* Body weight : ≥50.0 kg, <85.0 kg
* Body Mass Index : ≥17.6, <26.4
* Healthy, as judged by the investigator/subinvestigator based on the results of physical examinations (subjective symptoms and objective findings) and all tests obtained at screening and during the period from hospital admission in Period 1 to immediately before study medication

Exclusion Criteria:

* Subjects with the following history.

  1. Hepatic disease (e.g. viral hepatitis, drug-induced liver injury).
  2. Heart disease (e.g. congestive heart failure, angina pectoris, arrhythmia requiring

     treatment).
  3. Respiratory disease (e.g. serious bronchial asthma, chronic bronchitis)
  4. Gastrointestinal disease (e.g. serious peptic ulcer, gastroesophageal reflux esophagitis;

     diseases requiring several selections except for appendicitis)
  5. Renal disease (e.g. acute renal failure, glomerulonephritis, interstitial nephritis).
  6. Cerebrovascular disorder (e.g. cerebral infarction).
  7. Malignant tumor.
  8. Drug allergies. Allergic disorders (except for hay fever)
  9. Any use of drugs abuse. Alcohol abuse
* Any concurrent illness (except for caries)
* A deviation from the normal reference range of blood pressure, pulse rate, body temperature, or 12-lead ECG at screening or upon admission in Period 1 (day preceding the day of study medication).
* Any deviation of the following criteria for clinical laboratory tests at screening or upon admission in Period 1 (day preceding the day of study medication). The normal reference ranges specified at the study site will be used as the normal reference ranges in the present study.

  1. Hematology:

     * A deviation of ±20% from the upper or lower limit of the normal range
  2. Blood biochemistry:

     * A deviation from the normal range for AST, ALT, creatinine (Cre), or serum electrolytes.
     * A deviation of ±20% from the upper or lower limit of the normal range for other items than the above.
     * However, the lower limit of the normal range will not be established for items for which a deviation from the lower limit is not considered clinically significant[AST, ALT, total bilirubin (T-Bil), ALP, γ-GTP, LDH, CK, Cre, uric acid (UA)and total cholesterol (T-Cho)].
  3. Urinalysis:

     * U-Glu, U-Pro ≥+1
     * U-Uro ≥+2
  4. Urinary drug test: A positive result for phencyclidine, benzodiazepine, cocaine, amphetamines, cannabis, opiates, barbiturates or tricyclic antidepressants
  5. Immunological test: A positive result for HBs antigen, HCV antibody, syphilis, or HIV antigen/antibody
* Received medication within 14 days before hospital admission in Period 1 or is scheduled to receive medication
* Received any investigational drugs in other clinical or post-marketing studies within 120 days before the screening assessment
* Previous treatment with FK949E
* Donated more than 400 mL of whole blood within 90 days, more than 200 mL of whole blood within 30 days, or blood components within 14 days before the screening assessment
* Excessive smoking or drinking habit (measure of "excessive": alcohol: 45 g/day [a 633 mL bottle of beer contains 25 g of alcohol, and 180 mL of Japanese sake contains 22 g of alcohol], smoking: 20 cigarettes/day).
* Other subjects concerned ineligible by the investigator/subinvestigator

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of unchanged quetiapine | For 48 hours after dosing
AUC (area under the curve) of unchanged quetiapine | For 48 hours after dosing

SECONDARY OUTCOMES:
tmax of plasma concentration of unchanged quetiapine | For 48 hours after dosing
t1/2 of plasma concentration of unchanged quetiapine | For 48 hours after dosing
Safety assessed by the incidence of adverse events, clinical lab tests, vital signs, 12-lead ECGs and physical exam | Up to 48 hours after each administration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Kyushu, Japan

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=178